CLINICAL TRIAL: NCT01074216
Title: Vitamin D Levels in Stage IV Colorectal Cancer Patients: A Phase II Study
Brief Title: Vitamin D Levels in Stage IV Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-143
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Colorectal Cancer
Keywords: Vitamin D; Vitamin D3; colon cancer; rectum cancer; Cholecalciferol; 09-143
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cholecalciferol

ARMS (1):
- vitamin D, vitamin D3 (Experimental): This is a Phase II study involving Stage IV colorectal cancer patients with serum vitamin D deficiency, to determine the ability to correct vitamin D deficiency and to maintain serum vitamin D levels (25-hydroxy vitamin D) once achieved.
  Interventions: Drug: vitamin D repletion with Cholecalciferol (vitamin D3 50,000 International Units)

INTERVENTIONS:
Drug: vitamin D repletion with Cholecalciferol (vitamin D3 50,000 International Units) — Patients will be given vitamin D repletion with Cholecalciferol (vitamin D3 50,000 International Units) three times per week until the target vitamin D level of 40 ng/ml is achieved, and vitamin D3 maintenance initiated at 2,000 International Units daily thereafter.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, vitamin D blood levels has on stage IV colorectal cancer. Tbe doctors want to see if it is possible to increase low vitamin D levels into normal range using vitamin D supplements taken by mouth. Low vitamin D levels have been associated with worse outcomes in persons who have cancer. Low vitamin D may also cause people to have symptoms such as pain and fatigue. We want to see if increasing low vitamin D levels will help improve cancer outcomes. Vitamin D is routinely repleted in all subjects known to be vitamin D deficient. Therefore, the treatment given would be considered standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage IV (metastatic) colorectal cancer
* Baseline 25-hydroxy vitamin D level < 30 ng/ml
* Age ≥18 years of age

Exclusion Criteria:

* Current or previous malignancy except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for > 3 years
* Albumin < 3.2
* Patients on concurrent chronic steroids, other than those allowed for routine antiemetics, or inhaled steroids
* Patients receiving phenobarbital, phenytoin, orlistat and cholestyramine
* Hypercalcemia (Calcium >10.5 mg/dl)
* Calcium x Phosphorus > 70 mg2/dL2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Wesa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Stage IV colorectal cancer patients will be given vitamin D repletion with Cholecalciferol (vitamin D3 50,000 International Units) three times per week until the target vitamin D level of 40 ng/ml is achieved, and vitamin D3 maintenance initiated at 2,000 International Units daily thereafter.
Period: Overall Study
Arm/Group | All Patients
Started | 54
Completed | 41
Not Completed | 13
Not completed — Physician Decision | 1
Not completed — Not Treated | 12

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: To Achieve Target Vitamin D Level
Description: To determine the ability of achieving the target serum 25-hydroxy vitamin D level of 40 ng/ml within 6 weeks of beginning vitamin D supplements in patients with metastatic colon cancer. A response is defined as achieving serum vitamin D levels ≥40 ng/ml at least once at any point during the first 6 weeks
Time Frame: Within 6 weeks of beginning vitamin D
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 41
participants | 41

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 13/54
Other Adverse Events (participants affected / at risk) | 37/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=54)
Abdominal pain (General disorders) | 2 (2)
Allergic reaction (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (General disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (General disorders) | 1 (2)
Fever (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prostate infection (Infections and infestations) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Surgical and medical procedures - Other (General disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (3)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=54)
Abdominal pain (General disorders) | 8
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 6
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 9
Anorexia (General disorders) | 5
Anxiety (Psychiatric disorders) | 3
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 7
Blood bilirubin increased (Metabolism and nutrition disorders) | 8
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 14
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 9
Prothrombin ratio and international normalized ratio increased (Blood and lymphatic system disorders) | 7
Lymphocyte count decreased (Blood and lymphatic system disorders) | 8
Mucositis oral (General disorders) | 6
Neutrophil count decreased (Blood and lymphatic system disorders) | 14
Pain (General disorders) | 4
Pain in extremity (General disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 8
Platelet count decreased (Blood and lymphatic system disorders) | 6
Surgical and medical procedures - Other (General disorders) | 4
White blood cell decreased (Blood and lymphatic system disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes